CLINICAL TRIAL: NCT01853566
Title: Effects of Growth Hormone Administration on Muscle Strength and Body Composition in Men Over 50 Years Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Ana Beatriz Winter Tavares, Master degree in Endocrinology, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: GH and men
Record Dates: First submitted 2013-05-07; First posted 2013-05-15 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Muscle Strength; Growth Hormone; men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- growth hormone (Experimental): GH group received an initial dose of 0.5 units (UI)/day (0.2 mg/day), with readjustments to 1.0 UI/day (0.4 mg/day) and 1.5 UI/day (0.6 mg/day) after 1 and 2 months of treatment, respectively. The last GH dose will be maintained until the end of the study (6 months).
  Interventions: Drug: growth hormone

INTERVENTIONS:
Drug: growth hormone — GH group intervention: use of GH - initial dose of 0.5 UI/day (0.2 mg/day), with readjustments to 1.0 UI/day (0.4 mg/day) and 1.5 UI/day (0.6 mg/day) after 1 and 2 months of treatment, respectively. The last GH dose will be maintained until the end of the study. These GH dosages were based on the dose used for adults of the same age with GHD. Subjects will be re-evaluated after 6 months of GH therapy or placebo according to muscle strength and body composition .The other group received placebo using the same scheme as the GH group.
  Other Names: somatotropin

SUMMARY:
The growth hormone (GH) secretion declines gradually with age, with studies demonstrating a progressive reduction of 14% secretion per decade of life beginning in the second decade. Other studies suggest a disruption in GH secretion in elderly people. These findings suggest a possible association between growth hormone deficiency (GHD) and the ageing process.GH replacement is well known to improve body composition, leading to a decrease in total body fat and an increase in lean body mass. However, GH replacement has only shown an effect on muscle strength in GH-deficient adults subjected to long-term GH therapy. Few studies have evaluated the effect of GH replacement on muscle strength in elderly people engaged in a program of exercise training.Our purpose is to evaluate the effect of GH therapy on muscle strength in healthy, non-sedentary men over 50 years old.

DETAILED DESCRIPTION:
At baseline, subjects are submitted to evaluation of GH secretion, testosterone level, body composition, and muscle strength. Absence of GHD and normal testosterone levels were necessary for the inclusion in the study. These parameters will be evaluated after 6 months of GH use x placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and non-sedentary men aged 50-70 years

Exclusion Criteria:

* pituitary disease, GH use in the last 12 months, severe acute disease, hepatic and/or renal chronic disease, uncontrolled systemic arterial hypertension, diabetes mellitus, psychiatric disorders, history of cancer, non-treated hypogonadism and the presence of any other disease that could interfere with the somatotrophic axis.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Muscle strength after GH replacement | after 6 months of GH replacement
  Muscle strength is evaluated for the maximum strength based on the concept of maximum repetition (1 MR) (i.e., the maximum load that can be performed using the correct technique for an exercise).The exercises evaluated were bench press and leg press. To determine the load associated with 10 MR, each subject can initially performed 10 repetitions of each exercise with a sub maximum load, which is considered a load that was possible to mobilise. Then, the loads are progressively increased and with a maximum of 3 trials, the load of 10 MR is reached. During the 10 MR test, a 2-5 minute interval is provided between the attempts of each exercise. After the load was obtained for a determined exercise, intervals not less than 10 minutes were given before moving on to the next exercise.

SECONDARY OUTCOMES:
body composition after growth hormone replacement | after 6 months of growth hormone
  Body mass index is calculated using Quetelet's formula (weight/height2) and the percentage of body fat was calculated using the adipometer on seven cutaneous folds (tricipital, subscapular, suprailiac, pectoral, axillary, abdominal and thigh) according to the Pollock and Jackson protocol. Abdominal circumference is measured using a non-elastic tape at the greatest diameter between the last ribs and the iliac crests. The same person examined all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Beatriz tavares, Principal Investigator — Hospital Universitário Clementino Fraga Filho - UFRJ
Locations (1):
- Hospital Universitário Clementino Fraga Filho - UFRJ, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Tavares AB, Micmacher E, Biesek S, Assumpcao R, Redorat R, Veloso U, Vaisman M, Farinatti PT, Conceicao F. Effects of Growth Hormone Administration on Muscle Strength in Men over 50 Years Old. Int J Endocrinol. 2013;2013:942030. doi: 10.1155/2013/942030. Epub 2013 Dec 8. PMID 24382963